CLINICAL TRIAL: NCT03151798
Title: Nutrient Overload, Insulin Resistance, and Hepatic Mitochondrial Dysfunction
Brief Title: The Liver Health Study for Patients with NAFLD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Elizabeth Jane Parks, Professor, Nutrition and Exercise Physiology, University of Missouri-Columbia
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: 2008258
Record Dates: First submitted 2017-05-10; First posted 2017-05-12 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2023-07

CONDITIONS: Nonalcoholic Fatty Liver; Nonalcoholic Steatohepatitis; Obesity
Keywords: Nonalcoholic fatty liver; Exercise; Weight loss diet
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Obesity; Motor Activity

STUDY DESIGN:
Intervention Model Description: In Phase I, liver samples derived from patients undergoing either bariatric surgery or a liver biopsy to diagnose nonalcoholic fatty liver disease, are tested one time in vitro. There is no treatment in Phase I.
  In Phase II, only patients with nonalcoholic fatty liver disease (and not those who have had bariatric surgery) are eligible to go into a study in which they are randomly assigned to 1) a lifestyle treatment program or 2) a control group undergoing standard care. Allocation is 2:1 subjects in the treatment vs standard care groups.
  Thus, the arms are:
  Arm 1: Phase I studies with no treatment, only observational data generated in vitro from the liver samples Arm 2: Phase II lifestyle treatment Arm 3: Phase II control standard of care
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Phase I: Observational studies (Experimental): Patients are eligible who are undergoing either bariatric surgery or a liver biopsy for the diagnosis of nonalcoholic fatty liver disease
  Interventions: Other: Phase I: Observational studies
- Phase II: Lifestyle treatment (Experimental): Subjects will undergo lifestyle modification to cause weight loss and improved fitness
  Interventions: Behavioral: Phase II: Lifestyle treatment
- Phase II: Control treatment (Placebo Comparator): Subjects will be given dietary advice and a stretching program.
  Interventions: Behavioral: Phase II: Control treatment

INTERVENTIONS:
Behavioral: Phase II: Lifestyle treatment — Subjects will undergo energy restriction and exercise training over a 9 month period.
  Arms: Phase II: Lifestyle treatment
Behavioral: Phase II: Control treatment — Subjects will receive dietary advice and receive information on a stretching program.
  Arms: Phase II: Control treatment
Other: Phase I: Observational studies — The liver samples from patients undergoing bariatric surgery or a diagnostic liver biopsy will undergo in vitro assays to determine the capacity of the tissue to burn fat
  Arms: Phase I: Observational studies

SUMMARY:
The study will investigate whether the level of fat stored in the liver is related to the liver's ability to burn fat.

DETAILED DESCRIPTION:
The study has two phases. In Phase I, liver samples from patients undergoing bariatric surgery or a diagnostic liver biopsy will be tested for the ability to burn fatty acids. In Phase II, patients with nonalcoholic fatty liver disease will participate in either a nine-month lifestyle treatment program or undergo standard care. The goal is to determine how weight loss and exercise improve liver health.

Inpatient comprehensive metabolic tests are performed before and after the nine-months.

ELIGIBILITY:
For Phase I: Any patient scheduled to undergo bariatric surgery or a liver biopsy to diagnose nonalcoholic fatty liver disease.

For Phase II: Only subjects who have had a diagnosis of nonalcoholic fatty liver disease and completed Phase I (and no subjects who have undergone bariatric surgery)

Inclusion Criteria:

1. Men and women (pre and post-menopausal)
2. Overweight/obese with BMI ≥ 25.9 or < 50.0 kg/m2
3. Characteristics of the metabolic syndrome, pre-diabetes (fasting glucose 100-125 mg/dL or 2h glucose 140-200 mg/dL) or diabetes type 2, or undergoing bariatric surgery
4. 22-65 years of age
5. Sedentary, < 60 minutes per week of structured physical activity
6. Alcohol intake< 20 g/d

Exclusion Criteria:

1. Having undergone bariatric surgery.
2. Acute disease or advanced cardiac or renal disease, anticoagulation therapy, or any severe co-morbid condition limiting life expectancy < 1 years
3. Other causes of hepatitis including hepatitis B & C, autoimmune hepatitis, hemochromatosis, celiac disease, Wilson's disease, alpha-1-antitrypsin deficiency, medication-induced hepatitis, any clinical or biochemical evidence of decompensated liver disease
4. Use of steroids or other drugs that cause NAFLD
5. Pregnant or trying to become pregnant
6. Inability to exercise on a bike or treadmill

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Actual)
Dates: Start 2017-08-09 (Actual); Primary Completion 2022-03-03 (Actual); Study Completion 2023-04-29 (Actual)

PRIMARY OUTCOMES:
Liver mitochondrial gene expression | 1 day
  Liver tissue will be tested in vitro to determine the abundance of transcript indicative of fat oxidation.

SECONDARY OUTCOMES:
Liver mitochondrial fat oxidation | 1 day
  Liver tissue will be tested in vitro to determine its capacity to burn fat
Histology to determine the amount of fibrosis in the liver | 1 day
  Liver samples will be tested to determine the severity of liver disease and whether diet and exercise reduce liver fibrosis.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Parks, PhD, Principal Investigator — University of Missouri-Columbia; Jamal Ibdah, MD, Principal Investigator — University of Missouri-Columbia; Scott Rector, PhD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Syed-Abdul MM, Moore MP, Wheeler A, Ganga RR, Diaz-Arias A, Rector RS, Ibdah JA, Parks EJ. Improvements in nonalcoholic fatty liver disease (NAFLD) after metabolic surgery is linked to an increased hepatic fatty acid oxidation-a case report. AME Surg J. 2021 Jun 30;1:4. doi: 10.21037/asj-20-5. PMID 40255245
- [Derived] Mucinski JM, Salvador AF, Moore MP, Fordham TM, Anderson JM, Shryack G, Cunningham RP, Lastra G, Gaballah AH, Diaz-Arias A, Ibdah JA, Rector RS, Parks EJ. Histological improvements following energy restriction and exercise: The role of insulin resistance in resolution of MASH. J Hepatol. 2024 Nov;81(5):781-793. doi: 10.1016/j.jhep.2024.06.017. Epub 2024 Jun 22. PMID 38914313